CLINICAL TRIAL: NCT03424408
Title: Serum Thromboxane B2 Assay as a Measure of Platelet Production in Healthy Volunteers Taking Aspirin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Noel Chan, Assistant Professor, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3626
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Aspirin
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aspirin 81 mg (Other): Healthy volunteers will receive 5 days of aspirin. Following cessation of aspirin, daily blood samples will be collected for serum thromboxane B2 measurement
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Aspirin 81 mg — Healthy volunteers will receive 5 days of aspirin 81 mg daily. Following cessation of aspirin, daily blood samples will be collected for serum thromboxane B2 measurement
  Other Names: Aspirin

SUMMARY:
Some aspirin-treated patients have a blunted pharmacological response predisposing to clinical failure. The investigators hypothesize that the blunted response often results from increased rate of platelet production and some failures will be prevented by administering aspirin twice daily. The overall objective is to develop a valid method to quantify platelet production (without the use of radioactive isotopes) in order to examine the hypothesis that enhanced platelet production is a common cause of poor aspirin responsiveness in patients with atherothrombosis.

DETAILED DESCRIPTION:
The specific objective of this study is to validate the Cayman Chemical serum thromboxane immunoassay as a measure of platelet production in healthy subjects who are treated with aspirin by demonstrating that the recovery of their serum thromboxane B2 levels occurs at a rate of about 10% per day after aspirin cessation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smoking volunteers;
* Age ≥ 18 years;

Exclusion Criteria:

* Allergy or intolerance to aspirin;
* Current pregnancy;
* Use of aspirin or drugs interfering with platelet function (NSAIDs, anticoagulants) within one week of study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Serum thromboxane B2 | daily for 5 days after aspirin cessation
  The daily rate of platelet production can be estimated by calculating the daily recovery rate of serum thromboxane B2 after aspirin over 5 days following aspirin cessation for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Noel Chan, MBBS, Principal Investigator — Hamilton Health Science
Locations (1):
- Thrombosis and Atherosclerosis Research Institute. Hamilton General Site, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03424408/Prot_000.pdf